CLINICAL TRIAL: NCT00006044
Title: A Phase I Trial of Testosterone in Patients With Progressive Androgen-Independent Prostate Cancer
Brief Title: Testosterone in Treating Patients With Progressive Prostate Cancer That No Longer Responds to Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-115; P30CA008748 (NIH); P01CA005826 (NIH); MSKCC-99115; NCI-G00-1818
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Testosterone Propionate

INTERVENTIONS:
Drug: therapeutic testosterone

SUMMARY:
RATIONALE: High doses of testosterone may be effective in killing prostate cancer cells that no longer respond to hormone therapy.

PURPOSE: Phase I trial to study the effectiveness of testosterone in treating patients who have progressive prostate cancer that no longer responds to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and maximum tolerated dose of exogenously administered testosterone in patients with progressive androgen-independent prostate cancer who have been in castrate state either surgically or pharmacologically for a minimum of 1 year.
* Assess the changes in expression of androgen receptor and other receptors in human biopsy specimens or circulating tumor cells before and after this treatment in this patient population.

OUTLINE: This is a dose-escalation study.

Patients receive testosterone via an enhanced absorption transdermal system continuously for 28 days. The transdermal patches are changed daily.

Cohorts of 3-6 patients receive a fixed daily dose of testosterone with escalating duration of exposure until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicities.

Patients are followed at day 1 and at weeks 2 and 4.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed androgen independent metastatic prostate cancer
* Progressive disease manifested by either:

  * New osseous lesions by bone scan or a greater than 25% increase in bidimensionally measurable soft tissue disease or the appearance of new sites of disease by MRI or CT scan OR
  * Minimum of 3 rising PSA values from baseline that are obtained 1 week or more apart, or 2 rising PSA values more than 1 month apart, where the percentage increase over the range of values is at least 25%
* Castrate state by orchiectomy or gonadotropin-releasing hormone analogues for minimum of 1 year

  * Testosterone no greater than 30 ng/mL
* Measurable disease
* Metastatic disease by bone scan, MRI, or CT scan
* Rising PSA values
* If receiving antiandrogen therapy, must have shown progressive disease off treatment
* No active CNS or epidural tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT less than 3 times upper limit of normal
* PTT less than 14 seconds

Renal:

* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV cardiac disease

Pulmonary:

* No severe debilitating pulmonary disease

Other:

* No infection requiring IV antibiotics
* No other severe medical problems that would increase risk for toxicity

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior biologic therapy
* No concurrent immunotherapy

Chemotherapy:

* Recovered from prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* If no prior orchiectomy, must continue on gonadotropin-releasing hormone analogs to maintain castrate levels of testosterone
* No concurrent finasteride
* No other concurrent hormonal therapy

Radiotherapy:

* Recovered from prior radiotherapy
* No concurrent radiotherapy to an indicator lesion

Surgery:

* See Disease Characteristics
* Recovered from prior surgery
* No concurrent surgery on only measurable lesion

Other:

* At least 4 weeks since other prior investigational anticancer drugs and recovered
* No other concurrent investigational anticancer agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Morris MJ, Huang D, Kelly WK, Slovin SF, Stephenson RD, Eicher C, Delacruz A, Curley T, Schwartz LH, Scher HI. Phase 1 trial of high-dose exogenous testosterone in patients with castration-resistant metastatic prostate cancer. Eur Urol. 2009 Aug;56(2):237-44. doi: 10.1016/j.eururo.2009.03.073. Epub 2009 Apr 3. PMID 19375217